CLINICAL TRIAL: NCT05012631
Title: Losartan for Diffuse Myocardial Fibrosis in Sickle Cell Disease: A Prospective, Phase II Study.
Brief Title: Losartan for Diffuse Myocardial Fibrosis in Sickle Cell Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Losartan-CMR
Record Dates: First submitted 2021-07-15; First posted 2021-08-19 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Sickle Cell Disease; Diffuse Myocardial Fibrosis
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Losartan

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Losartan (Experimental): Participants will receive oral losartan as tablets or oral solution one time daily. The dosing will depend on age and will be based on drug label and dosing used in studies on patients with SCD.
  Interventions: Drug: Losartan

INTERVENTIONS:
Drug: Losartan — Losartan dosing for participants <16 years will be 0.7 mg/kg (maximum of 50 mg) once daily. The dose can be increased to 1.4 mg/kg (maximum of 100 mg once daily) after 2 weeks if the dose was tolerated (no hypotension or hyperkalemia). For patients ≥16 years, the starting dose will be 50 mg once daily which can be increased to 100 mg daily if tolerated after 2 weeks.

SUMMARY:
This study is a pilot, phase II, open-label study of the angiotensin II receptor blocker, losartan, in patients with Sickle Cell Disease (SCD) 6 years or older for 12 months. The investigators will enroll 24 patients with SCD over the course of 1 year with a goal to complete all study procedures in 2 years. The short-term goal is to obtain clinical pilot data regarding the safety and efficacy of losartan in stabilizing or decreasing extracellular volume fraction (ECV) after 12 months of therapy.

ELIGIBILITY:
Inclusion Criteria:

1. 6 years old or older
2. Diagnosis of HbSS or Sbeta0-thalassemia
3. Ability to cooperate with and undergo CMR without sedation or anesthesia
4. Ability to cooperate with and undergo echocardiogram without sedation or anesthesia
5. Patients who are on a stable dose of sickle cell disease-modifying therapy: Hydroxyurea, Voxelotor, L-Glutamine, or Crizanlizumab, for 3 months prior to enrollment will be eligible.

Exclusion Criteria:

1. Current chronic transfusion therapy. Patients who received a simple transfusion for an acute event will be eligible 3 months after completion of transfusion
2. SCD genotypes other than specified in inclusion criteria
3. Any contraindication to CMR such as metallic implants
4. Inability to cooperate with CMR or echocardiography imaging
5. Known congenital heart disease
6. Estimated GFR ≤ to 30 mL/min/1.73 m2 by creatinine clearance
7. Pregnant or lactating females or females of child-bearing potential who are unable to use a medically accepted form of contraception throughout the study
8. Treatment with a renin-angiotensin pathway inhibitor during the 2 weeks prior to enrollment
9. Hypersensitivity to angiotensin receptor II blockers
10. Hyperkalemia (K>5.5 mEq/L) on a non-hemolyzed sample despite low-potassium diet
11. Hepatic dysfunction defined as serum ALT > 5x the upper normal limit for age
12. Current lithium therapy
13. Chronic daily use of NSAID
14. HIV infection.

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in extracellular volume fraction (ECV) after 1 year of losartan treatment | after 1 year of losartan treatment.
  Efficacy of losartan in stabilizing or reducing ECV (diffuse myocardial fibrosis) in SCD after one year.

SECONDARY OUTCOMES:
Change in Diastolic Function | after 1 year of losartan treatment.
  Efficacy of losartan in improving diastolic function defined by echocardiographic and tissue Doppler assessment .
Change in Exercise Capacity | after 1 year of losartan treatment.
  Efficacy of losartan in improving cardiopulmonary exercise testing (CPET) measurements.
Predicting Myocardial Fibrosis | At baseline and after one year of losartan treaement
  Explore the performance characteristics of the following serum biomarkers in predicting myocardial fibrosis in patients with SCD: PICP, PIIINP, TGF-β, CTGF, soluble ST2, galectin-3, and NT-proBNP.

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No